CLINICAL TRIAL: NCT00595647
Title: BAsel Stent Kosten Effektivitäts Trial - SAphenous Venous Graft Angioplasty Using Glycoprotein IIb/IIIa Receptor Inhibitors and Drug-Eluting Stents
Brief Title: Study to Test the Efficacy and Safety of Drug Eluting vs. Bare-Metal Stents for Saphenous Vein Graft Interventions
Acronym: BASKET-SAVAGE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Leipzig (Other)
Responsible Party: Principal Investigator, Raban Jeger, PD Dr. med. / MD, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASKET-SAVAGE EKBB# 278/07; SNF 3200B0_120029 (Other Grant/Funding Number: Schweizer Nationalfond); EKBB 278/07 (Other: Ethics Committee)
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Percutaneous coronary intervention
  Interventions: Device: Drug eluting stent
- 2 (Placebo Comparator): Percutaneous coronary intervention
  Interventions: Device: Bare metal stent

INTERVENTIONS:
Device: Drug eluting stent — Implantation of stent
  Other Names: TAXUS Liberté
  Arms: 1
Device: Bare metal stent — Implantation of stent
  Other Names: Liberté
  Arms: 2

SUMMARY:
Prospective multicenter controlled randomized trial to compare the safety and efficacy of drug eluting vs. bare metal stents in percutaneous coronary interventions of saphenous vein grafts. Hypothesis: Survival and outcome will be significantly better in patients receiving DES than in patients receiving BMS regarding both short-term and long-term outcome.

DETAILED DESCRIPTION:
Research Question: What is the effect of the paclitaxel eluting TAXUS® Liberté® stent compared with the bare-metal Liberté® stent (both Boston Scientific Corporation, Natick, MA) in saphenous vein graft (SVG) percutaneous coronary interventions (PCI) when used in conjunction with a glycoprotein IIb/IIIa inhibitor, e.g., abciximab (ReoPro®, Eli Lilly & Co., Indianapolis, IN), and a distal filter system? Design: Prospective, multicenter, controlled randomized trial. Subjects: Inclusion criteria: Patients undergoing SVG PCI with a target vessel reference diameter ≤ 5.5 mm (visual estimate); documented silent ischemia, stable angina pectoris Canadian Cardiovascular Society (CCS) class I to IV, or acute coronary syndrome. Exclusion criteria: Previous stent implantation anywhere in the target SVG; concomitant native vessel PCI; SVG age <6 months; arterial grafts; oral anticoagulation; platelet count <100x109/L or >700x109/L; any major non-cardiac condition with a life expectancy <12 months; known allergies against the components tested; white blood cell count <3000 cell/mm3; enrolled in other study; no consent; patients unlikely to comply to the study treatment and the follow-up visits. Recruitment: Consecutive sample of all patients who qualify Variables: Predictor: Randomization will be single-blinded 1:1 to the TAXUS® Liberté® vs. the Liberté® stent (both Boston Scientific Corporation, Natick, MA). In all patients, a distal filter system will be used during PCI. The use of a glycoprotein IIb/IIIa inhibitor, e.g., abciximab (ReoPro®, Eli Lilly & Co., Indianapolis, IN), will be strongly recommended (bolus prior to PCI and 12 h infusion post PCI). Outcome: Primary: MACE after 12 months. MACE will be defined as the composite of cardiac death (all deaths not clearly non-cardiac), non-fatal myocardial infarction, and TVR. Secondary: Non-fatal myocardial infarction and cardiac death at 30 days and 6, 12, 36, and 60 months; MACE at 30 days and 6, 36, and 60 months; quality of life; individual components of the primary endpoint; non-cardiac death; major bleeding, defined as need for surgery, need for blood transfusions, and cerebral hemorrhage during antiplatelet therapy; minor bleeding, defined as a drop in hematocrit of >2 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing SVG PCI with a target vessel reference diameter ≤ 5.5 mm (visual estimate)
* Documented silent ischemia, stable angina pectoris Canadian Cardiovascular Society (CCS) class I to IV, or acute coronary syndrome

Exclusion Criteria:

* Previous stent implantation anywhere in the target SVG
* Concomitant native vessel PCI
* SVG age <6 months
* Arterial grafts
* Oral anticoagulation
* Platelet count <100x109/L or >700x109/L, white blood cell count <3000 cells/mm3
* Any major non-cardiac condition with a life expectancy <12 months
* Planned elective surgery in the next 12 months
* Known allergies against the components tested
* Enrolled in other study
* No consent
* Patients unlikely to comply to the study treatment and the follow-up visits
* Age <18 years
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2008-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
MACE (composite of cardiac death, i.e., all deaths not clearly non-cardiac, non-fatal myocardial infarction, and TVR | 12 months

SECONDARY OUTCOMES:
Non-fatal MI and cardiac death; MACE; QoL; individual components of the primary endpoint; non-cardiac death; major bleeding; minor bleeding | 30 days and 6, 12, 36, and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Pfisterer, MD, Principal Investigator — University Hospital, Basel, Switzerland; Raban Jeger, MD, Principal Investigator — University Hospital, Basel, Switzerland; Sven Möbius-Winkler, MD, Principal Investigator — University of Leipzig/Heart Center, Germany
Locations (5):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Hellerup
- University of Leipzig/Heart Center, Leipzig, Germany
- Switzerland (2):
  - University Hospital Basel, Basel
  - Triemli Hospital, Zurich

REFERENCES:
- [Derived] Fahrni G, Farah A, Engstrom T, Galatius S, Eberli F, Rickenbacher P, Conen D, Mueller C, Pfister O, Twerenbold R, Coslovsky M, Cattaneo M, Kaiser C, Mangner N, Schuler G, Pfisterer M, Mobius-Winkler S, Jeger RV; BASKET-SAVAGE-Investigators*. Long-Term Results After Drug-Eluting Versus Bare-Metal Stent Implantation in Saphenous Vein Grafts: Randomized Controlled Trial. J Am Heart Assoc. 2020 Oct 20;9(20):e017434. doi: 10.1161/JAHA.120.017434. Epub 2020 Oct 9. PMID 33032485